CLINICAL TRIAL: NCT06358833
Title: Comparison of Postoperative Pain When Using an Endodontic Needle and Endo1 Ultrasonic Endo Activate Device During Root Canal Irrigation: A Randomized Controlled Pragmatic Clinical Trial
Brief Title: Comparison of Endodontic Postoperative Pain Using Different Irrigation Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Muhammad Zubair Ahmad, Associate Professor, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-82-03
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain; Irreversible Pulpitis
Keywords: root canal treatment; irrigation; ultrasonic activation; Endo1 Ultrasonic Endo Activate Device
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be masked from the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endodontic needle (EN) (Active Comparator): In this group, the irrigation of root canals will be done with 2.5 % sodium hypochlorite. The delivery of the irrigant will be done using 27G side-vented endodontic irrigation needles (Omega, Inc). The tip of the needle will be pre-measured and positioned within 1 millimeter of the working length. No activation of the irrigant will be performed.
  Interventions: Procedure: endodontic needle (EN)
- Endodontic activation (EA) (Experimental): In this group, the irrigation of root canals will be done with 2.5% sodium hypochlorite. The delivery of the irrigant will be done using 27G side-vented endodontic irrigation needles (Omega, Inc). The irrigant will be activated with ultrasonic energy using the Endo-1 Ultrasonic Endo Activator (Guilin Woodpecker, Guilin, China). The tip of the Endo-1 Ultrasonic Endo Activator device will be pre-measured and kept within 1 mm from the working length. The manufacturer's instructions regarding irrigant activation will be followed.
  Interventions: Procedure: Endodontic activation (EA)

INTERVENTIONS:
Procedure: endodontic needle (EN) — the irrigation of root canals will be done with 2.5 % sodium hypochlorite. The delivery of the irrigant will be done using 27G side-vented endodontic irrigation needles (Omega, Inc). The tip of the needle will be pre-measured and positioned within 1 millimeter of the working length. No activation of the irrigant will be performed.
  Arms: Endodontic needle (EN)
Procedure: Endodontic activation (EA) — the irrigation of root canals will be done with 2.5% sodium hypochlorite. The delivery of the irrigant will be done using 27G side-vented endodontic irrigation needles (Omega, Inc). The irrigant will be activated with ultrasonic energy using the Endo-1 Ultrasonic Endo Activator (Guilin Woodpecker, Guilin, China). The tip of the Endo-1 Ultrasonic Endo Activator device will be pre-measured and kept within 1 mm from the working length. The manufacturer's instructions regarding irrigant activation will be followed.
  Arms: Endodontic activation (EA)

SUMMARY:
Summary:

After a root canal procedure, it is common to experience postoperative pain. Cleaning the root canal thoroughly is crucial for pain relief, but removing all debris with standard methods is difficult. Irrigation, using either traditional endodontic needles or newer methods like endodontic activation, helps clean the canal. This study aims to compare pain levels after using conventional needles versus an Endo1 Ultrasonic Endo Activate Device for irrigation. Patients will undergo standard root canal preparation and then be randomly assigned to one of two groups for final irrigation: the Endo1 device (EA) and the conventional endodontic needles (EN). The study will provide insights into which method is more effective in reducing postoperative pain.

DETAILED DESCRIPTION:
Background:

One of the primary objectives following root canal therapy is to alleviate pain. While postoperative pain is undesirable, it is often considered a common sensation following endodontic treatment.

Completely removing all organic and inorganic debris from the root canal system to ensure the elimination of irritants that can cause postoperative pain is a challenging task, even when using precise rotary, hand, or hybrid instruments. Therefore, irrigation plays a crucial role in the cleaning and shaping process.

Traditional root canal irrigation typically involves the use of an endodontic needle (EN) to disinfect the root canal. However, a newer approach called endodontic activation (EA) has been suggested to enhance root canal disinfection by activating irrigants within the canal.

Both of these methods of root canal irrigation are routine practice and part of the standard root canal treatment.

Rationale:

No study has directly compared the effects of final irrigation using conventional endodontic needles and an Endo1 Ultrasonic Endo Activate Device (Guilin Woodpecker, Guilin, China) on postoperative pain using a pragmatic approach. Therefore, the objective of this study is to assess and compare postoperative pain following the utilization of closed-ended endodontic needles and the Endo1 Ultrasonic Endo Activate Device during final root canal irrigation.

Study objectives:

The study aims to assess and compare the levels of postoperative pain following endodontic activation (EA) of irrigants using the Endo1 Ultrasonic Endo Activate Device (Guilin Woodpecker, Guilin, China) versus conventional endodontic needle (EN) irrigation in root canal therapy.

Methods In this prospective single-blind, parallel-armed, randomized clinical trial, standard root canal preparation will be done; patients will be randomly assigned into one of the two groups. In the final irrigation protocol, group EA will go through activation using Endo1 Ultrasonic Endo Activate Device while patients in group EN will receive irrigation by conventional endodontic needle technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) visiting the College of Dentistry and undergoing root canal treatment in posterior teeth (molars and premolars).
* Teeth having fully formed roots with mature apices.
* Patients willing to collaborate in the study must sign a written consent form.
* Diagnosis of irreversible pulpitis in posterior tooth/teeth requiring root canal treatment.
* No history of allergy to the anesthesia solution.
* Classified as class I, II in the American Society of Anesthesiologists Physical Status Classification System.

Exclusion Criteria:

* Patients diagnosed with pulp necrosis in the tooth require root canal treatment.
* Mentally or medically compromised patients.
* Pregnant women.
* Patients on any medications for the past two weeks
* Patients who refuse to participate in the study.
* Patients with a history of allergy from any of the contents of local anesthesia or rubber dam material.
* Non-restorable teeth

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 6 hours postoperatively
  Postoperative pain will be measured using the Heft-Parker visual analog scale (VAS)
Postoperative pain | 12 hours postoperatively
  Postoperative pain will be measured using the Heft-Parker visual analog scale (VAS)
Postoperative pain | 48 hours postoperatively
  Postoperative pain will be measured using the Heft-Parker visual analog scale (VAS)
Postoperative pain | 1 week postoperatively
  Postoperative pain will be measured using the Heft-Parker visual analog scale (VAS)

SECONDARY OUTCOMES:
Irrigation time | During root canal treatment
  Time spent in irrigation procedures

OTHER OUTCOMES:
Adverse event | During and immediately after root canal treatment
  If any adverse event will occur, it will be recorded
Rescue medication | Up-to 1 week postoperatively
  In case of unbearable postoperative pain, the principal investigator will prescribe oral analgesic (ibuprofen 200 mg as the over-the-counter drug), and the timepoint of medication intake will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Zubair Ahmad, FCPS, Principal Investigator — Qassim University, Saudi Arabia
Locations (1):
- Muhammad Zubair Ahmad, Ar Rass, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of IPD is subjected to further approval from the Committee of Research Ethics, the institutional review board (IRB) of Qassim University.